CLINICAL TRIAL: NCT07302152
Title: Evaluation of Elastosonographic Techniques Implemented on Ultrasound Systems for the Assessment of Liver Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Gianluigi Poma, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: p_12
Record Dates: First submitted 2025-11-26; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-02

CONDITIONS: Liver Stiffness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Age > 18 years cohort (Other)
  Interventions: Diagnostic Test: elastosonographic

INTERVENTIONS:
Diagnostic Test: elastosonographic — Measurement performed in the right intercostal space, using the median value of 5 measurements for 2D shear wave and 10 measurements for point shear wave

SUMMARY:
The assessment of liver stiffness is essential in patients with suspected or confirmed chronic liver disease, as clinical management depends on the degree and progression of hepatic fibrosis, which increases liver hardness. In recent years, non-invasive elastosonographic techniques have been introduced to estimate liver fibrosis. The first to be implemented was Transient Elastography (TE), which has shown high accuracy in identifying significant fibrosis and cirrhosis, particularly in patients with HCV-related chronic liver disease, and has been endorsed by The European Association for the Study of the Liver (EASL) guidelines as an alternative to liver biopsy. More recently, shear-wave elastography techniques integrated into conventional ultrasound systems have been developed, offering the advantage of real-time B-mode ultrasound guidance. The aim of this study is to compare these techniques with each other and with TE.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, ability to hold breath during image acquisition, informed consent.

Exclusion Criteria:

* any condition that, in the investigator's clinical judgment, would make further participation in the study unacceptable for that individual patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
elastosonographic | up to 24 months
  Measurement taken in the right intercostal space, median value of 5 measurements for 2D shear wave and 10 measurements for point shear wave.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SSD Malattie Infettive 3 - Ecografia, Pavia, Pavia, Italy